CLINICAL TRIAL: NCT01370642
Title: A Phase III Randomized, Placebo-controlled Study to Evaluate the Safety, Tolerability, and Efficacy of MK-7009 When Administered Concomitantly With Peginterferon Alfa-2b and Ribavirin in Japanese Treatment-Naïve Patients With Chronic Hepatitis C Infection
Brief Title: Vaniprevir Administered With Pegylated-interferon and Ribavirin in Japanese Treatment-Naïve Chronic Hepatitis C Participants (MK-7009-043)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7009-043
Record Dates: First submitted 2011-06-08; First posted 2011-06-10 (Estimated); Results first posted 2014-10-06 (Estimated); Last update posted 2018-10-18 (Actual); Status verified 2018-09

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — vaniprevir; peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Vaniprevir 12 Week Arm (Experimental): Participants on this arm receive 12 weeks of vaniprevir (300 mg twice daily) and then 12 weeks of placebo to vaniprevir along with 24 weeks of treatment with peg-IFN and RBV.
  Interventions: Drug: vaniprevir; Drug: Placebo to vaniprevir; Biological: Peg-IFN; Drug: ribavirin
- Vaniprevir 24 Week Arm (Experimental): Participants on this arm receive 24 weeks of vaniprevir (300 mg twice daily) along with 24 weeks of treatment with peg-IFN and RBV.
  Interventions: Drug: vaniprevir; Biological: Peg-IFN; Drug: ribavirin
- Control Arm (Active Comparator): Participants on this arm receive 24 weeks of treatment with placebo to vaniprevir along with 48 weeks of treatment with peg-IFN and RBV.
  Interventions: Drug: Placebo to vaniprevir; Biological: Peg-IFN; Drug: ribavirin

INTERVENTIONS:
Drug: vaniprevir — Capsules containing 150 mg vaniprevir, orally, two in the morning and two in the evening for 12 or 24 weeks
  Other Names: MK-7009
  Arms: Vaniprevir 12 Week Arm; Vaniprevir 24 Week Arm
Drug: Placebo to vaniprevir — Placebo to vaniprevir, capsules, orally, twice daily for 12 weeks or 24 weeks
  Arms: Control Arm; Vaniprevir 12 Week Arm
Biological: Peg-IFN — Peg-IFN 1.5 μg/kg once per week, subcutaneously (SC) for 24 or 48 weeks
  Other Names: PegIntron
Drug: ribavirin — Capsules containing 200 mg RBV orally, 3 to 5 capsules, dosage based on the participant's weight (600 mg/day to 1000 mg/day), for 24 or 48 weeks
  Other Names: REBETOL®

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and efficacy of vaniprevir given in combination with pegylated interferon alfa-2b (peg-IFN) and ribavirin (RBV) versus treatment with peg-IFN and RBV alone in Japanese treatment-naïve participants with chronic hepatitis C (CHC) genotype (GT)1. The primary efficacy hypothesis is that the percentage of participants achieving sustained virologic response 24 weeks after completion of all study therapy (SVR24) in at least one of the vaniprevir arms is superior to the percentage of participants achieving SVR24 in the control arm.

ELIGIBILITY:
Inclusion criteria:

* Japanese participant diagnosed with compensated CHC GT 1
* Absence of ascites, bleeding esophageal varices, hepatic encephalopathy, or other signs or symptoms of advanced liver disease.
* IFN treatment naive
* No evidence of cirrhosis

Exclusion criteria:

* Co-infection with human immunodeficiency virus (HIV)
* Positive hepatitis B surface antigen or other evidence of active hepatitis B infection
* Any other condition that is contraindicated or for which caution is required for treatment with peg-IFN or RBV
* Any condition or pre-study laboratory abnormality, or history of any illness, that, in the opinion of the investigator, might confound the results of the study or pose additional risk in administering the study drugs, peg-IFN and RBV, to the participant.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Actual)
Dates: Start 2011-06-27 (Actual); Primary Completion 2013-07-31 (Actual); Study Completion 2014-03-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Hayashi N, Nakamuta M, Takehara T, Kumada H, Takase A, Howe AY, Ludmerer SW, Mobashery N. Vaniprevir plus peginterferon alfa-2b and ribavirin in treatment-naive Japanese patients with hepatitis C virus genotype 1 infection: a randomized phase III study. J Gastroenterol. 2016 Apr;51(4):390-403. doi: 10.1007/s00535-015-1120-x. Epub 2015 Sep 25. PMID 26403160
- [Derived] Ludmerer SW, Hirano T, Black S, Howe AY, Chang W, Takase A, Nakamura K, Tanaka Y, Kumada H, Hayashi N, Nickle D. HCV evolutionary genetics of SVR versus virologic failure assessed from the vaniprevir phase III registration trials. Antiviral Res. 2016 Jun;130:118-29. doi: 10.1016/j.antiviral.2016.03.004. Epub 2016 Mar 3. PMID 26947564
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=7009-043&kw=7009-043&tab=access

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Japanese patients 20-70 years old (inclusive) who had chronic, compensated, genotype 1 Hepatitis C (HCV) infection, and HCV ribonucleic acid (RNA) levels ≥ 5.0 log IU/mL peripheral blood at screening were recruited from 55 sites in Japan.
Pre-assignment Details: Of 294 randomized participants, 293 received at least 1 dose of study treatment and comprised the All Participants As Treated Population (APaT) as well as the Full Analysis Set (FAS). One treated participant was excluded from the FAS and APaT due to a protocol violation.
Period: Overall Study
Arm/Group | Vaniprevir 12 Week Arm | Vaniprevir 24 Week Arm | Control Arm
Started | 98 | 98 | 98
FAS Population | 98 | 97 | 98
Completed | 90 | 92 | 69
Not Completed | 8 | 6 | 29
Not completed — Adverse Event | 2 | 1 | 1
Not completed — Detectable HCV RNA | 0 | 0 | 22
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Physician Decision | 4 | 1 | 2
Not completed — Withdrawal by Subject | 2 | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vaniprevir 12 Week Arm | Vaniprevir 24 Week Arm | Control Arm | Total
Number analyzed (Participants) | 98 | 98 | 98 | 294
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.2 (12.0) | 55.5 (9.7) | 54.8 (9.9) | 54.5 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 49 | 52 | 157
  Male | 42 | 49 | 46 | 137

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Sustained Virologic Response 24 Weeks After Completion of All Study Therapy (SVR24)
Description: SVR24 was defined as having an undetectable HCV RNA level 24 weeks after completion of all study therapy.
Time Frame: 24 weeks after 24 or 48 weeks of study therapy (up to 72 weeks)
Population: Full Analysis Set (FAS) population; all randomized participants who received at least one dose of study treatment. One treated participant was excluded from the FAS due to a protocol violation.
Measure: Number; unit: percentage of participants
Arm/Group | Vaniprevir 12 Week Arm | Vaniprevir 24 Week Arm | Control Arm
Number analyzed (Participants) | 98 | 97 | 98
percentage of participants | 83.7 | 84.5 | 55.1
Statistical Analysis 1: Comparison: Vaniprevir 12 Week Arm vs Control Arm; To compare the percentage of participants achieving SVR24 between the vaniprevir and control arms, 95% confidence intervals and corresponding p-values for the between-treatment difference (vaniprevir - control) were computed using Miettinen and Nurminen method stratified by Interleukin 28B (IL28B) and age utilizing Cochran-Mantel-Haenszel weights; Test type: Superiority or Other; p < 0.001, Miettinen and Nurminen method; Adjusted Difference in Percentages = 29.0, 95% CI 2-sided [17.2 to 40.5]
Statistical Analysis 2: Comparison: Vaniprevir 24 Week Arm vs Control Arm; To compare the percentage of participants achieving SVR24 between the vaniprevir and control arms, 95% confidence intervals and corresponding p-values for the between-treatment difference (vaniprevir - control) were computed using Miettinen and Nurminen method stratified by IL28B and age utilizing Cochran-Mantel-Haenszel weights; Test type: Superiority or Other; p < 0.001, Miettinen and Nurminen method; Adjusted Difference in Percentages = 28.6, 95% CI 2-sided [17.4 to 40.0]

2. Secondary Outcome: Percentage of Participants Achieving SVR12
Description: SVR12 was defined as having an undetectable HCV RNA level 12 weeks after completion of all study therapy.
Time Frame: 12 weeks after 24 or 48 weeks of study therapy (up to 60 weeks)
Population: FAS population; all randomized participants who received at least one dose of study treatment. One treated participant was excluded from the FAS due to a protocol violation.
Measure: Number; unit: percentage of participants
Arm/Group | Vaniprevir 12 Week Arm | Vaniprevir 24 Week Arm | Control Arm
Number analyzed (Participants) | 98 | 97 | 98
percentage of participants | 83.7 | 84.5 | 54.1
Statistical Analysis 1: Comparison: Vaniprevir 12 Week Arm vs Control Arm; To compare the percentage of participants achieving SVR12 between the vaniprevir and control arms, 95% confidence intervals and corresponding p-values for the between-treatment difference (vaniprevir - control) were computed using Miettinen and Nurminen method stratified by IL28B and age utilizing Cochran-Mantel-Haenszel weights; Test type: Superiority or Other; p < 0.001, Miettinen and Nurminen method; Adjusted Difference in Percentages = 30.0, 95% CI 2-sided [18.1 to 41.5]
Statistical Analysis 2: Comparison: Vaniprevir 24 Week Arm vs Control Arm; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Miettinen and Nurminen method; Adjusted Difference in Percentages = 29.6, 95% CI 2-sided [18.3 to 41.0]

3. Secondary Outcome: Percentage of Participants Achieving Rapid Virologic Response (RVR)
Description: RVR was defined as having an undetectable HCV RNA level at Week 4.
Time Frame: At Week 4
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Vaniprevir 12 Week Arm | Vaniprevir 24 Week Arm | Control Arm
Number analyzed (Participants) | 98 | 97 | 98
percentage of participants | 86.7 | 85.6 | 9.2
Statistical Analysis 1: Comparison: Vaniprevir 12 Week Arm vs Control Arm; To compare the percentage of participants achieving RVR between the vaniprevir and control arms, 95% confidence intervals and corresponding p-values for the between-treatment difference (vaniprevir - control) were computed using Miettinen and Nurminen method stratified by IL28B and age utilizing Cochran-Mantel-Haenszel weights; Test type: Superiority or Other; p < 0.001, Miettinen and Nurminen method; Adjusted Difference in Percentages = 78.1, 95% CI 2-sided [68.2 to 85.3]
Statistical Analysis 2: Comparison: Vaniprevir 24 Week Arm vs Control Arm; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.001, Miettinen and Nurminen method; Adjusted Difference in Percentages = 76.7, 95% CI 2-sided [66.7 to 84.1]

4. Secondary Outcome: Percentage of Participants Achieving Complete Early Virologic Response (cEVR)
Description: cEVR was defined as having an undetectable HCV RNA level at Week 12.
Time Frame: At Week 12
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Vaniprevir 12 Week Arm | Vaniprevir 24 Week Arm | Control Arm
Number analyzed (Participants) | 98 | 97 | 98
percentage of participants | 94.9 | 96.9 | 46.9
Statistical Analysis 1: Comparison: Vaniprevir 12 Week Arm vs Control Arm; To compare the percentage of participants achieving cEVR between the vaniprevir and control arms, 95% confidence intervals and corresponding p-values for the between-treatment difference (vaniprevir - control) were computed using Miettinen and Nurminen method stratified by IL28B and age utilizing Cochran-Mantel-Haenszel weights; Test type: Superiority or Other; p < 0.001, Miettinen and Nurminen method; Adjusted Difference in Percentages = 48.4, 95% CI 2-sided [37.2 to 58.9]
Statistical Analysis 2: Comparison: Vaniprevir 24 Week Arm vs Control Arm; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, Miettinen and Nurminen method; Adjusted Difference in Percentages = 49.6, 95% CI 2-sided [38.5 to 60.0]

5. Secondary Outcome: Percentage of Participants Achieving Undetectable HCV RNA at the End of Treatment (EOT)
Description: Participants were assessed for undetectable HCV RNA levels at the end of all study therapy.
Time Frame: At Week 24 or 48
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Vaniprevir 12 Week Arm | Vaniprevir 24 Week Arm | Control Arm
Number analyzed (Participants) | 98 | 97 | 98
percentage of participants | 95.9 | 97.9 | 79.6
Statistical Analysis 1: Comparison: Vaniprevir 12 Week Arm vs Control Arm; To compare the percentage of participants achieving undetectable HCV RNA at EOT between the vaniprevir and control arms, 95% confidence intervals and corresponding p-values for the between-treatment difference (vaniprevir - control) were computed using Miettinen and Nurminen method stratified by IL28B and age utilizing Cochran-Mantel-Haenszel weights; Test type: Superiority or Other; p < 0.001, Miettinen and Nurminen method; Adjusted Difference in Percentages = 17.0, 95% CI 2-sided [8.1 to 27.3]
Statistical Analysis 2: Comparison: Vaniprevir 24 Week Arm vs Control Arm; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.001, Miettinen and Nurminen method; Adjusted Difference in Percentages = 17.8, 95% CI 2-sided [9.3 to 27.8]

6. Primary Outcome: Percentage of Participants With One or More Tier 1 Adverse Events (AEs) During the Study
Description: An adverse experience was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which is temporally associated with the use of the product, was also an adverse experience. For this study, safety parameters or AEs of special interest that were identified a priori constituted "Tier 1" safety endpoints that were subject to inferential testing for statistical significance. Tier 1 AEs on this study included serious rash, anemia (anemia plus haemoglobin decreased), neutropenia (neutropenia plus neutrophil count decreased), bilirubin increased and gastrointestinal adverse (GI) experiences (vomiting, nausea, and diarrhea).
Time Frame: From Day 1 (post-dose) through completion of Week 24 Follow-up (up to 72 weeks)
Population: All Participants Treated (APaT) Population; all participants receiving at least one dose of study treatment. One treated participant was excluded from the APaT due to a protocol violation.
Measure: Number; unit: percentage of participants
Arm/Group | Vaniprevir 12 Week Arm | Vaniprevir 24 Week Arm | Control Arm
Number analyzed (Participants) | 98 | 97 | 98
percentage of participants
  With ≥1 Tier 1 AEs | 89.8 | 83.5 | 85.7
  anaemia | 60.2 | 51.5 | 64.3
  bilirubin increased | 7.1 | 12.4 | 701
  GI AEs | 62.2 | 52.6 | 46.9
  neutropenia | 59.2 | 51.5 | 51.0
Statistical Analysis 1: Comparison: Vaniprevir 12 Week Arm vs Control Arm; Difference in percentage of participants with ≥1 Tier 1 AEs between vaniprevir and control; Test type: Superiority or Other; p = 0.385, Miettinen and Nurminen method; Difference in percentages = 4.1, 95% CI 2-sided [-5.4 to 13.7]
Statistical Analysis 2: Comparison: Vaniprevir 24 Week Arm vs Control Arm; Difference in percentage of participants with ≥1 Tier 1 AEs between vaniprevir and control; Test type: Superiority or Other; p = 0.670, Miettinen and Nurminen method; Difference in percentages = -2.2, 95% CI 2-sided [-12.6 to 8.1]
Statistical Analysis 3: Comparison: Vaniprevir 12 Week Arm vs Control Arm; Difference in percentage of participants with anemia Tier 1 AEs between vaniprevir and control; Test type: Superiority or Other; p = 0.557, Miettinen and Nurminen method; Difference in percentages = -4.1, 95% CI 2-sided [-17.5 to 9.5]
Statistical Analysis 4: Comparison: Vaniprevir 24 Week Arm vs Control Arm; Difference in percentage of participants with anemia Tier 1 AEs between vaniprevir and control; Test type: Superiority or Other; p = 0.072, Miettinen and Nurminen method; Difference in percentages = -12.7, 95% CI 2-sided [-26.2 to 1.2]
Statistical Analysis 5: Comparison: Vaniprevir 12 Week Arm vs Control Arm; Difference in percentage of participants with bilirubin increased Tier 1 AEs between vaniprevir and control; Test type: Superiority or Other; p > 0.999, Miettinen and Nurminen method; Difference in percentages = 0.0, 95% CI 2-sided [-7.9 to 7.9]
Statistical Analysis 6: Comparison: Vaniprevir 24 Week Arm vs Control Arm; Difference in percentage of participants with bilirubin increased Tier 1 AEs between vaniprevir and control; Test type: Superiority or Other; p = 0.220, Miettinen and Nurminen method; Difference in percentages = 5.2, 95% CI 2-sided [-3.3 to 14.2]
Statistical Analysis 7: Comparison: Vaniprevir 12 Week Arm vs Control Arm; Difference in percentage of participants with GI Tier 1 AEs between vaniprevir and control; Test type: Superiority or Other; p = 0.032, Miettinen and Nurminen method; Difference in percentages = 15.3, 95% CI 2-sided [1.3 to 28.7]
Statistical Analysis 8: Comparison: Vaniprevir 24 Week Arm vs Control Arm; Difference in percentage of participants with GI Tier 1 AEs between vaniprevir and control; Test type: Superiority or Other; p = 0.432, Miettinen and Nurminen method; Difference in percentages = 5.6, 95% CI 2-sided [-8.4 to 19.4]
Statistical Analysis 9: Comparison: Vaniprevir 12 Week Arm vs Control Arm; Difference in percentage of participants with neutropenia Tier 1 AEs between vaniprevir and control; Test type: Superiority or Other; p = 0.252, Miettinen and Nurminen method; Difference in percentages = 8.2, 95% CI 2-sided [-5.8 to 21.8]
Statistical Analysis 10: Comparison: Vaniprevir 24 Week Arm vs Control Arm; Difference in percentage of participants with neutropenia Tier 1 AEs between vaniprevir and control; Test type: Superiority or Other; p = 0.942, Miettinen and Nurminen method; Difference in percentages = 0.5, 95% CI 2-sided [-13.4 to 14.4]

7. Secondary Outcome: Least Squares (LS) Mean Change From Baseline in HCV RNA (Log 10)
Description: HCV RNA levels were assessed at baseline (BL) and during treatment weeks 2, 4, 8, 12, and 24 using the Roche TaqMan HCV assay, and transformed to Log 10 values. HCV RNA values below the limit of reliable quantification (LoQ) or the limit of detection (LoD) at any time point were handled as follows (imputations done for computational purposes): values below the LoQ but above the LoD were imputed with the LoQ minus 0.1; values below the LoD were imputed with the value of 0 Log IU/mL. HCV RNA levels below the LoD were considered "undetectable".
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12, Week 24
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Log IU/ml
Arm/Group | Vaniprevir 12 Week Arm | Vaniprevir 24 Week Arm | Control Arm
Number analyzed (Participants) | 98 | 97 | 98
Log IU/ml
  Change From BL at Week 2 | -5.3 [-5.5 to -5.1] | -5.5 [-5.7 to -5.3] | -2.0 [-2.2 to -1.8]
  Change From BL at Week 4 | -6.0 [-6.3 to -5.8] | -6.1 [-6.3 to -5.9] | -3.0 [-3.3 to -2.8]
  Change From BL at Week 8 | -6.1 [-6.4 to -5.9] | -6.2 [-6.4 to -5.9] | -4.2 [-4.5 to -4.0]
  Change From BL at Week 12 | -6.1 [-6.4 to -5.9] | -6.2 [-6.4 to -5.9] | -4.8 [-5.0 to -4.5]
  Change From BL at Week 24 | -6.0 [-6.3 to -5.8] | -6.1 [-6.4 to -5.9] | -5.3 [-5.5 to -5.0]
Statistical Analysis 1: Comparison: Vaniprevir 12 Week Arm vs Control Arm; Change from BL in HCV RNA at Week 2 was computed using a constrained longitudinal data analysis model including treatment, time and the interaction of time by treatment with a restriction of the same baseline mean across treatment groups as well as adjusting for IL28B and age, and their interaction terms with time will be included in the model; Test type: Superiority or Other; Constrained LDA Model; LS Mean Difference at Week 2 = -3.2, 95% CI 2-sided [-3.5 to -3.0]
Statistical Analysis 2: Comparison: Vaniprevir 24 Week Arm vs Control Arm; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; Constrained LDA Model; LS Mean Difference at Week 2 = -3.5, 95% CI 2-sided [-3.7 to -3.2]
Statistical Analysis 3: Comparison: Vaniprevir 12 Week Arm vs Control Arm; Change from BL in HCV RNA at Week 4 was computed using a constrained longitudinal data analysis model including treatment, time and the interaction of time by treatment with a restriction of the same baseline mean across treatment groups as well as adjusting for IL28B and age, and their interaction terms with time will be included in the model; Test type: Superiority or Other; Constrained LDA Model; LS Mean Difference at Week 4 = -3.0, 95% CI 2-sided [-3.3 to -2.7]
Statistical Analysis 4: Comparison: Vaniprevir 24 Week Arm vs Control Arm; [analysis description as in outcome 7, analysis 3]; Test type: Superiority or Other; Constrained LDA Model; LS Mean Difference at Week 4 = -3.1, 95% CI 2-sided [-3.4 to -2.8]
Statistical Analysis 5: Comparison: Vaniprevir 12 Week Arm vs Control Arm; Change from BL in HCV RNA at Week 8 was computed using a constrained longitudinal data analysis model including treatment, time and the interaction of time by treatment with a restriction of the same baseline mean across treatment groups as well as adjusting for IL28B and age, and their interaction terms with time will be included in the model; Test type: Superiority or Other; Constrained LDA Model; LS Mean Difference at Week 8 = -1.9, 95% CI 2-sided [-2.2 to -1.6]
Statistical Analysis 6: Comparison: Vaniprevir 24 Week Arm vs Control Arm; [analysis description as in outcome 7, analysis 5]; Test type: Superiority or Other; Constrained LDA Model; LS Mean Difference at Week 8 = -2.0, 95% CI 2-sided [-2.3 to -1.7]
Statistical Analysis 7: Comparison: Vaniprevir 12 Week Arm vs Control Arm; Change from BL in HCV RNA at Week 12 was computed using a constrained longitudinal data analysis model including treatment, time and the interaction of time by treatment with a restriction of the same baseline mean across treatment groups as well as adjusting for IL28B and age, and their interaction terms with time will be included in the model; Test type: Superiority or Other; Constrained LDA Model; LS Mean Difference at Week 12 = -1.4, 95% CI 2-sided [-1.7 to -1.1]
Statistical Analysis 8: Comparison: Vaniprevir 24 Week Arm vs Control Arm; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; Constrained LDA Model; LS Mean Difference at Week 12 = -1.4, 95% CI 2-sided [-1.7 to -1.1]
Statistical Analysis 9: Comparison: Vaniprevir 12 Week Arm vs Control Arm; Change from BL in HCV RNA at Week 24 was computed using a constrained longitudinal data analysis model including treatment, time and the interaction of time by treatment with a restriction of the same baseline mean across treatment groups as well as adjusting for IL28B and age, and their interaction terms with time will be included in the model; Test type: Superiority or Other; Constrained LDA Model; LS Mean Difference at Week 24 = -0.8, 95% CI 2-sided [-1.1 to -0.5]
Statistical Analysis 10: Comparison: Vaniprevir 24 Week Arm vs Control Arm; [analysis description as in outcome 7, analysis 9]; Test type: Superiority or Other; Constrained LDA Model; LS Mean Difference at Week 24 = -0.9, 95% CI 2-sided [-1.2 to -0.6]

8. Primary Outcome: Percentage of Participants Who Discontinued Study Drug Due to an AE
Description: An adverse experience was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which is temporally associated with the use of the product, was also an adverse experience.
Time Frame: From Day 1 (post-dose) through completion of Week 24 Follow-up (up to 72 weeks)
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Vaniprevir 12 Week Arm | Vaniprevir 24 Week Arm | Control Arm
Number analyzed (Participants) | 98 | 97 | 98
percentage of participants | 7.1 | 3.1 | 11.2

ADVERSE EVENTS:
Time Frame: From Day 1 (post-dose) through completion of Week 24 Follow-up (up to 72 weeks)
Description: AEs reported for APaT population. AEs were not reported for one participant in the Vaniprevir 24 Week Arm.
Arm/Group | Vaniprevir 12 Week Arm | Vaniprevir 24 Week Arm | Control Arm
Serious Adverse Events (participants affected / at risk) | 5/98 | 6/97 | 9/98
Other Adverse Events (participants affected / at risk) | 98/98 | 97/97 | 98/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vaniprevir 12 Week Arm (N=98) | Vaniprevir 24 Week Arm (N=97) | Control Arm (N=98)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Endolymphatic hydrops (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Sudden hearing loss (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Heat stroke (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Ligament injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Glycosylated haemoglobin increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vaniprevir 12 Week Arm (N=98) | Vaniprevir 24 Week Arm (N=97) | Control Arm (N=98)
Anaemia (Blood and lymphatic system disorders) | 25 (26) | 19 (19) | 22 (24)
Neutropenia (Blood and lymphatic system disorders) | 8 (10) | 4 (4) | 7 (8)
Vertigo (Ear and labyrinth disorders) | 3 (4) | 3 (3) | 5 (7)
Dry eye (Eye disorders) | 7 (7) | 7 (7) | 2 (2)
Retinal haemorrhage (Eye disorders) | 1 (1) | 1 (1) | 6 (6)
Retinopathy (Eye disorders) | 3 (3) | 7 (7) | 12 (12)
Abdominal discomfort (Gastrointestinal disorders) | 16 (19) | 18 (20) | 10 (13)
Abdominal pain upper (Gastrointestinal disorders) | 12 (14) | 10 (10) | 8 (10)
Cheilitis (Gastrointestinal disorders) | 6 (6) | 7 (7) | 4 (4)
Constipation (Gastrointestinal disorders) | 11 (12) | 12 (13) | 11 (12)
Dental caries (Gastrointestinal disorders) | 2 (2) | 5 (6) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 30 (32) | 21 (25) | 22 (31)
Dyspepsia (Gastrointestinal disorders) | 13 (14) | 7 (7) | 6 (6)
Gastritis (Gastrointestinal disorders) | 1 (1) | 6 (6) | 4 (4)
Nausea (Gastrointestinal disorders) | 36 (39) | 32 (38) | 27 (29)
Stomatitis (Gastrointestinal disorders) | 12 (13) | 29 (32) | 22 (25)
Vomiting (Gastrointestinal disorders) | 24 (29) | 30 (40) | 9 (10)
Chills (General disorders) | 1 (1) | 6 (6) | 1 (1)
Fatigue (General disorders) | 28 (31) | 29 (29) | 19 (21)
Influenza like illness (General disorders) | 6 (8) | 10 (10) | 12 (13)
Injection site erythema (General disorders) | 11 (12) | 14 (14) | 16 (17)
Injection site pruritus (General disorders) | 4 (4) | 8 (8) | 9 (10)
Injection site reaction (General disorders) | 24 (24) | 26 (26) | 28 (28)
Malaise (General disorders) | 31 (33) | 32 (33) | 37 (41)
Pyrexia (General disorders) | 79 (91) | 69 (108) | 80 (135)
Hepatic function abnormal (Hepatobiliary disorders) | 6 (6) | 3 (3) | 4 (4)
Cystitis (Infections and infestations) | 6 (6) | 3 (4) | 3 (3)
Nasopharyngitis (Infections and infestations) | 21 (27) | 29 (33) | 31 (42)
Accidental overdose (Injury, poisoning and procedural complications) | 2 (2) | 3 (3) | 6 (9)
Alanine aminotransferase increased (Investigations) | 2 (2) | 7 (7) | 7 (8)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 6 (6) | 7 (8)
Bilirubin conjugated increased (Investigations) | 2 (2) | 5 (5) | 2 (2)
Blood albumin decreased (Investigations) | 2 (2) | 5 (5) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 4 (4) | 6 (6) | 8 (8)
Blood bilirubin increased (Investigations) | 7 (7) | 12 (12) | 7 (7)
Blood calcium decreased (Investigations) | 7 (7) | 10 (11) | 6 (6)
Blood lactate dehydrogenase increased (Investigations) | 7 (11) | 6 (7) | 6 (7)
Blood phosphorus decreased (Investigations) | 5 (6) | 3 (3) | 5 (6)
Blood thyroid stimulating hormone increased (Investigations) | 2 (2) | 3 (3) | 11 (11)
Blood uric acid increased (Investigations) | 8 (8) | 5 (5) | 5 (5)
Gamma-glutamyltransferase increased (Investigations) | 6 (6) | 9 (9) | 11 (12)
Haematocrit decreased (Investigations) | 8 (8) | 2 (2) | 3 (3)
Haemoglobin decreased (Investigations) | 35 (37) | 31 (32) | 42 (49)
Lymphocyte count decreased (Investigations) | 5 (6) | 3 (3) | 2 (2)
Neutrophil count decreased (Investigations) | 50 (57) | 46 (50) | 43 (54)
Platelet count decreased (Investigations) | 28 (29) | 36 (36) | 36 (36)
Red blood cell count decreased (Investigations) | 7 (7) | 7 (7) | 7 (7)
Weight decreased (Investigations) | 15 (15) | 12 (12) | 9 (9)
White blood cell count decreased (Investigations) | 45 (47) | 44 (46) | 45 (45)
Decreased appetite (Metabolism and nutrition disorders) | 31 (32) | 32 (33) | 35 (36)
Arthralgia (Musculoskeletal and connective tissue disorders) | 30 (32) | 34 (35) | 29 (31)
Back pain (Musculoskeletal and connective tissue disorders) | 15 (15) | 17 (18) | 18 (18)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 3 (3) | 6 (7) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 9 (10) | 17 (18) | 12 (12)
Dizziness (Nervous system disorders) | 8 (9) | 6 (6) | 13 (14)
Dysgeusia (Nervous system disorders) | 26 (26) | 23 (23) | 19 (19)
Headache (Nervous system disorders) | 49 (55) | 47 (62) | 46 (59)
Insomnia (Psychiatric disorders) | 14 (15) | 23 (23) | 20 (20)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 11 (12) | 14 (15)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (3) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 11 (12) | 10 (12)
Alopecia (Skin and subcutaneous tissue disorders) | 31 (31) | 30 (30) | 33 (33)
Dry skin (Skin and subcutaneous tissue disorders) | 5 (5) | 7 (7) | 5 (5)
Eczema (Skin and subcutaneous tissue disorders) | 8 (9) | 4 (4) | 12 (14)
Erythema (Skin and subcutaneous tissue disorders) | 6 (6) | 5 (6) | 6 (7)
Pruritus (Skin and subcutaneous tissue disorders) | 29 (29) | 34 (35) | 35 (36)
Rash (Skin and subcutaneous tissue disorders) | 42 (45) | 33 (41) | 45 (50)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission.